CLINICAL TRIAL: NCT04869956
Title: Gut Microbiome Modification Through Dietary Intervention in Patients With Colorectal Cancer: Response to Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-2-7-HCUVA
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer
Keywords: Microbiome; Surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fatty Acids, Unsaturated

STUDY DESIGN:
Intervention Model Description: open, controlled, randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard diet (Other): Dietary pattern: Standard diet
  Interventions: Other: Dietary pattern: Standard diet
- High - Fiber diet rich in PUFA (Experimental): High - Fiber diet rich in PUFA
  Interventions: Other: Dietary pattern : High-fiber diet rich in PUFA

INTERVENTIONS:
Other: Dietary pattern : High-fiber diet rich in PUFA — High-fiber diet rich in PUFAs (total dietary intake of at least 30 grams of fiber per day, and of at least 3 grams of PUFAs per day from food, not supplements) at least 4 weeks before surgery
  Arms: High - Fiber diet rich in PUFA
Other: Dietary pattern: Standard diet — standard nutritional recommendations
  Arms: Standard diet

SUMMARY:
The investigators will conduct an open, controlled, randomized clinical trial, in patients with scheduled surgical intervention for CRC in the General Surgery and Digestive System Unit of the Virgen de la Arrixaca University Hospital (Murcia, Spain). All the included individuals must have passed the protocol of the Virgen de la Arrixaca University Hospital to be candidates for elective major surgery for CRC and must sign the informed consent after being informed of the objectives and the methodology of the study. The Helsinki Declaration will be followed during the duration of the project.

Patients will be randomized in a 1:1 ratio after receiving a diagnosis of CRC in the endoscopic evaluation; in the control arm, patients will receive standard nutritional recommendations, while patients in the intervention arm will be advised to follow a high-fiber diet rich in PUFAs (total dietary intake of at least 30 grams of fiber per day, and of at least 3 grams of PUFAs per day from food, not supplements) at least 4 weeks before surgery

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years old.
* After clinical diagnosis of CRC (stage I-III), the doctor has recommended and arranged for CRC surgery

Exclusion Criteria:

* Clinical diagnosis of stage IV CRC.
* Current gastrointestinal illness other than gastroesophageal reflux disease or hemorrhoids (such as celiac disease, inflammatory bowel disease, malabsorptive bariatric procedures, etc.).
* Chronic liver or kidney disease.
* History of cardiac disease.
* Positive genetic test for inherited polyposis syndromes (such as familial adenomatous polyps, hereditary non-polyposis colon cancer syndromes, etc).
* Alcoholism or illicit drug use.
* Antibiotic use within the past 2 months.
* Dietary supplement use including pre- or probiotics within the past month.
* History of intestinal cancer, inflammatory bowel disease, celiac disease, or malabsorptive bariatric surgery.
* Inflammatory or connective tissue disease (such as lupus, scleroderma, rheumatoid arthritis, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of anastomotic leakage | 360 Days from Baseline
  Number of anastomotic leakage
Surgical site infection | 360 Days from Baseline
  Number of site infection

SECONDARY OUTCOMES:
Change in gut microbiome composition | 360 Days from Baseline
  changes in gut microbiota composition by 16S rRNA gene sequencing
Serum levels of inflammation markers | 360 Days from Baseline
  Blood samples will be used to determine markers of inflammation (IL-6, IL-1β, IL-10 and TNFα), and markers of intestinal permeability (zonulin)
Length of hospitalization after surgery | 360 Days from Baseline
  Number of days
Recurrences of CRC after surgery | 360 Days from Baseline
  Number of recurrences

CONTACTS AND LOCATIONS:
Locations (1):
- Biomedical Research Institute of Murcia (IMIB-Arrixaca), Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided